CLINICAL TRIAL: NCT05185817
Title: Evaluation of COVID-19 Vaccine Effectiveness and Immunogenicity in Patients Receiving Hematopoietic Stem Cell Transplantation
Brief Title: Effectiveness of COVID-19 Vaccine in Hematopoietic Stem Cell Transplant Patients
Acronym: ESCVHSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1400-2-101-54534
Record Dates: First submitted 2022-01-10; First posted 2022-01-11 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2021-10

CONDITIONS: Hematopoietic Stem Cell Transplantation (HSCT); COVID-19 Vaccines; Immune System Tolerance
Keywords: hematopoietic stem cell transplantation, SARS-CoV-2 specific IgG , immune reconstitution, COVID-19 vaccine efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vaccine (Experimental): Patients who are a candidate for HSCT within the the Hematology, Oncology, and Stem Cell Transplantation Research Center of Shariaty Hospital, and agree to be vaccinated with an approved vaccine against the COVID-19 virus.
  Interventions: Biological: Pasocovac vaccine

INTERVENTIONS:
Biological: Pasocovac vaccine — All enrolled post-Allo-SCT participants who meet the inclusion criteria are recruited to study from 3 to 12 months after Allo-HSCT and vaccinated with 2 doses of Pastucovac, with a 4-week (±7 days) interval and a booster dose at an 8-week (±7 days) interval from the second dose.

SUMMARY:
COVID-19 vaccinations are predicted to be a huge success in pandemic control. However, the majority of the studies were conducted on healthy individuals, and the efficiency of COVID-19 vaccination in post-transplant patients is uncertain. In the setting of HSCT, the extreme immunosuppression caused by the conditioning regimen and the graft versus host disease (GvHD) preventive regimen clearly has an impact on the efficacy and immunogenicity of the COVID-19 vaccine. Given the importance of eliciting early SARS-Cov-2 protective immunity in patients who are undergoing Allo-HSCT and the EBMT recommendation to endorse vaccination as early as 3 months after allo-HCT [7], we conduct this prospective study to investigate the safety and immunogenicity of three doses Pastucovac (an RBD-based SARS-Cov-2 vaccine) at the early post-transplant period in adult Iranian patients who are undergoing Allo-HSCT. We also want to see whether there are any possible predictors, such as the effect of clinical characteristics and lymphocyte subpopulations at the time of vaccination on the serologic response following immunization. The findings of this study will serve to guide future COVID-19 vaccination recommendations in this population, such as the optimal starting time, interval time, and so on.

DETAILED DESCRIPTION:
From the start of the study until the sample size of 100 patients is attained, all consecutive adult patients who are candidates for Allo-SCT at HORCSCT, sign a research project consent to administer SARS-CoV-2 vaccination with Pastucovac, and sign a permission to take pre-and post-vaccination blood samples for deposit to the research database, are enrolled in the study. At baseline (before conditioning) and day +30 post-transplant, peripheral blood samples are taken to test particular lymphocyte subpopulations and SARS-CoV-2 IgG titers.

All enrolled post-Allo-SCT participants who meet the inclusion criteria including; age ≥ 18 years, successfully engraftment with full donor chimerism, absence of grade 3,4 acute GvHD or severe extensive chronic GvHD, no receive more than 0.5 mg/kg prednisolone, and no positive RT-PCR test for COVID-19 following HSCT are recruited to study from 3 to 12 months after Allo-HSCT and vaccinated with 2 doses of Pastucovac, with a 4-week (±7 days) interval and a booster dose with an 8-week (±7 days) interval from the second dose. Peripheral blood samples are collected before the first dose of vaccine to assess certain immune reconstitution and SARS-CoV-2 IgG titer. The serologic response against the SARS-CoV-2 spike protein (anti-S) is assessed in serum four weeks (± one week) after the first vaccine dose (before the second vaccine), four weeks (± one week) after the second dose, and four weeks (± one week) after the booster dose (third dose).

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years, successfully engraftment with full donor chimerism, absence of grade 3,4 acute GvHD or severe extensive chronic GvHD, no receive more than 0.5 mg/kg prednisolone, and no positive RT-PCR test for COVID-19 following HSCT

Exclusion Criteria:

Patients who are not candidates for the COVID-19 vaccine after transplantation due to severe complications.

Patients who do not consent to vaccination after transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of COVID-19 vaccine effectiveness | 4 weeks (±7 days) post second COVID-19 vaccine
  defined as a rising ≥ 4-fold in SARS-CoV-2 binding antibody titer compared to the pre-vaccine titer
Grade III-IV vaccine-related adverse reactions | 14 days after administration of each vaccine dose
  Prevalence of reactogenicity, Serious Adverse Events (SAE), and Suspected Unexpected Serious Adverse Reaction (SUSAR)

SECONDARY OUTCOMES:
Incidence of Acute Graft versus host disease (GvHD) | 4-week (±7 days) after second and third (booster) dose of vaccine.
  Measuring how the acute GvHD affect the response to the vaccine
GvHD prophylactic strategy affect immunological response | 4-week (±7 days) after third (booster) dose of vaccine.
  Measuring how early prophylactic immuno-suppression tapering affect the response to the vaccine
Immune cells recovery predicting the response to the COVID-19 vaccine | 4-week (±7 days) after third (booster) dose of vaccine.
  Measuring how early post HSCT Immune subsets reconstitution including T cells, NK cells, and B cells predict the seroconversion after second dose of vaccine.
seroconversion after second dose of vaccine | 4-week (±7 days) after second dose of vaccine.
  defined as a rising ≥ 4-fold in SARS-CoV-2 binding antibody titer compared to the pre-vaccine titer in patients starting their vaccination course 3-6 months after HSCT
seroconversion after second dose of vaccine | 4-week (±7 days) after second dose of vaccine.
  defined as a rising ≥ 4-fold in SARS-CoV-2 binding antibody titer compared to the pre-vaccine titer in patients starting their vaccination course 6-12 months after HSCT.
seroconversion after first dose of vaccine | 4-week (±7 days) after first dose of vaccine.
  defined as a rising ≥ 4-fold in SARS-CoV-2 binding antibody titer compared to the pre-vaccine titer
seroconversion after third (booster) dose of vaccine | 4-week (±7 days) after third (booster) dose of vaccine.
  defined as a rising ≥ 4-fold in SARS-CoV-2 binding antibody titer compared to the pre-vaccine titer
Incidence and severity of COVID-19 infections | 6 months following start of immunization
  Determine incidence and severity of COVID-19 infections by 6 months following immunization with a SARS-CoV-2 vaccine.
Correlation of seroconversion with patient characteristics | 4-week (±7 days) after second and third (booster) dose of vaccine.
  Determine how the patients characteristics including age, sex, performance score, and underlying disease affect on seroconversion

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Barkhordar, MD, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Hematology, Oncology, and Stem Cell Transplantation Research Center of shariaty Hospital, Tehran, Iran